CLINICAL TRIAL: NCT06698276
Title: Clinical and Histological Assessment of a Bone Substitute Enriched With Bioactive Glass for Ridge Preservation
Brief Title: Performance of Next-X in Alveolar Ridge Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Giuseppe Alexandre Romito, Chairman of Periodontics Division, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Next-X
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hopeless Tooth
Keywords: prospective case series

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2 months reopen group (Experimental): a biomaterial will be used to alveolar ridge preservation, and after 2 months participants of this group will receive a dental implant
  Interventions: Other: Alveolar Ridge Reconstruction
- 3 months reopen group (Experimental): a biomaterial will be used to alveolar ridge preservation, and after 3 months participants of this group will receive a dental implant
  Interventions: Other: Alveolar Ridge Reconstruction

INTERVENTIONS:
Other: Alveolar Ridge Reconstruction — It will be used a combination of two biomaterials for alveolar ridge preservation

SUMMARY:
The goal of this case series study is to evaluate the clinical and histological outcomes of a protocol for managing hopeless teeth, focusing on alveolar preservation and subsequent dental implant placement. The study will also assess the long-term success of prosthetic reconstruction. The main questions it aims to answer are:

* How effective is the use of biomaterials for alveolar preservation in maintaining bone structure and quality?
* What are the histological characteristics of the alveolar bone after biomaterial application?
* How successful are dental implants and prosthetic reconstructions in restored sites over a 1-year follow-up period?

Participants will:

1. Undergo extraction of hopeless teeth using an atraumatic protocol.
2. Receive alveolar preservation treatment with biomaterials immediately after extraction.
3. Provide a bone biopsy for histological processing before implant placement.
4. Undergo dental implant placement and prosthetic reconstruction of the lost tooth.
5. Attend follow-up appointments over a 1-year period for clinical and radiographic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 80 years of age.
* Requirement for single-rooted tooth extraction due to reasons such as caries, fractures, restorative issues, endodontic complications (e.g., root fracture, instrument fracture), orthodontic needs, or prosthetic considerations.
* Presence of at least one neighboring tooth adjacent to the extraction site.
* Maintaining adequate oral hygiene, indicated by bleeding on probing <20% and plaque index <20%.
* Presence of at least 50% of the buccal bone plate.
* Classification of patients as ASA I or II status according to the American Society of Anesthesiologists Classification.

Exclusion Criteria:

* All smokers, including smoking alternatives.
* Heavy drinker (> 60 g of alcohol per day as a mean).
* Uncontrolled metabolic disorders e.g., diabetes mellitus, osteomalacia, thyroid disorder, severe renal or hepatic disorder.
* Prolonged corticosteroid therapy.
* Immunological impairment diseases.
* History of malignancy, radiotherapy, or chemotherapy for malignancy within the past five years.
* General contraindications for dental and/or surgical treatment (including patients who take anticoagulants or antiresorptives).
* Disease or condition affecting bone metabolism.
* Women of child-bearing age, not using a highly effective method of birth control.
* Pregnancy or breast feeding.
* Previous and concurrent medication affecting sinus healing in general (e.g., topical steroids, large doses of anti-inflammatory drugs).
* Acute or chronic oral infection or uncontrolled periodontal disease.
* Crestal bone defects at the implantation site, which require additional bone augmentation around the neck of the implant.
* Allergy to collagen.
* Participation in an investigational device or drug clinical trial within the last six month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
histological analysis | Samples will be collected at 2 and 3 months after the surgical intervention
  Histological sections will be stained with hematoxylin-eosin (HE) and Masson's trichrome. A semi-quantitative analysis will be performed by a pathologist (Blinded for the groups), adopting a histological score system (0 - absence, 1- mild; 2 - mild to moderate, 3 - moderate to intense, and 4 - intense). These scores will be determined based on the intensity of the following histological parameters: necrosis, inflammatory infiltrate, fibrosis, biomaterial remnants, new-formed bone trabeculae, and angiogenesis. A histomorphometric analysis will also be performed for the trabecular bone area, cellularity area, and microvessel density.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Odontologia da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data can not be shared without he/she approval.